CLINICAL TRIAL: NCT03474744
Title: Copanlisib and Rituximab in Marginal Zone Lymphoma Patients (COUP-1)
Brief Title: Copanlisib and Rituximab in Marginal Zone Lymphoma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Buske (Other)
Collaborators: University of Ulm (Other); Optimapharm (Industry); X-act Cologne Clinical Research GmbH (Industry); Zentrum für Klinische Studien Ulm (Other); Celltrion Healthcare Co., LTD (Unknown); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Christian Buske, Prof. Dr. med., University of Ulm
Organization: University of Ulm (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COUP-1
Record Dates: First submitted 2018-02-28; First posted 2018-03-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Marginal Zone Lymphoma
Keywords: Copanlisib; Rituximab; Oncology
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Neoplasms | interventions — copanlisib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): Induction Phase:
  Cycle 1-6 (28 days cycle):
  Copanlisib: 60 mg i.v. fixed dose days 1, 8, 15. Rituximab: 375 mg/m2 day 1 i.v.
  Maintenance:
  Start 2 months after start of the last induction cycle for patients at least achieving a stable response after induction.
  Copanlisib: 60 mg i.v. fixed dose day 1 and day 15 every 4 weeks for a maximum of 12 cycles or until progression or study drug-related intolerable toxicity (month 2 to month 13 after end of induction).
  Rituximab: 375 mg/m2 i.v. day 1 every 8 weeks for a maximum of 12 infusions or until progression or study drug-related intolerable toxicity (month 2 to month 24 after end of induction)
  Interventions: Drug: Copanlisib; Drug: Rituximab

INTERVENTIONS:
Drug: Copanlisib — Solution for IV infusion
  Other Names: Aliqopa
Drug: Rituximab — Solution for IV infusion
  Other Names: Truxima

SUMMARY:
For marginal zone lymphoma (MZL) Rituximab in combination with conventional chemotherapy is widely used for those patients who fail local therapy or do not qualify for such. Depending on the MZL subtype Rituximab/chemotherapy is able to induce in part long remissions, but do not prevent relapse later on. In addition, chemotherapy associated toxicity is often problematic in MZL patients, who are mostly of advanced age. Thus, chemotherapy - free approaches are highly attractive for this patient group. Rituximab single agent is a widely used chemotherapy - free approach in MZL, but was significantly inferior compared to Rituximab/chlorambucil in a large randomized prospective clinical trial in treatment naïve MZL with a CR rate of 56 % vs. 80%, respectively (P<0.001). Thus, it is the major aim to develop chemotherapy - free approaches for MZL, which approach efficacy of Rituximab/chemotherapy combinations, but avoid chemotherapy associated toxicities. This in particular important in MZL as many physicians are reluctant to treat these often elderly patients with more intense treatments and prefer single agent therapies in these very often well and long responding lymphoma subtype. The PI3K inhibitor Copanlisib has shown high clinical activity in indolent B - cell lymphomas among them MZL. Based on these observations it is the aim of this study to test the toxicity and efficacy of Copanlisib in combination with the anti-CD20 antibody Rituximab in patients with newly diagnosed or relapsed MZL in need of treatment, who are not eligible or failed local therapy, following the assumption that this novel chemotherapy - free combination is significantly more effective than Rituximab single agent therapy and at least as efficient as Rituximab/chemotherapy, but avoids chemotherapy - related toxicity.

DETAILED DESCRIPTION:
For marginal zone lymphoma (MZL) Rituximab in combination with conventional chemotherapy is widely used for those patients who fail local therapy or do not qualify for such. Depending on the MZL subtype Rituximab/chemotherapy is able to induce in part long remissions, but do not prevent relapse later on. In addition, chemotherapy associated toxicity is often problematic in MZL patients, who are mostly of advanced age. Thus, chemotherapy - free approaches are highly attractive for this patient group. Rituximab single agent is a widely used chemotherapy - free approach in MZL, but was significantly inferior compared to Rituximab/chlorambucil in a large randomized prospective clinical trial in treatment naïve MZL with a CR rate of 56 % vs. 80%, respectively (P<0.001). Thus, it is the major aim to develop chemotherapy - free approaches for MZL, which approach efficacy of Rituximab/chemotherapy combinations, but avoid chemotherapy associated toxicities. This in particular important in MZL as many physicians are reluctant to treat these often elderly patients with more intense treatments and prefer single agent therapies in these very often well and long responding lymphoma subtype. The PI3K inhibitor Copanlisib has shown high clinical activity in indolent B - cell lymphomas among them MZL. Based on these observations it is the aim of this study to test the toxicity and efficacy of Copanlisib in combination with the anti-CD20 antibody Rituximab in patients with newly diagnosed or relapsed MZL in need of treatment, who are not eligible or failed local therapy, following the assumption that this novel chemotherapy - free combination is significantly more effective than Rituximab single agent therapy and at least as efficient as Rituximab/chemotherapy, but avoids chemotherapy - related toxicity.

The objective of the trial is to test the efficacy and toxicity of the treatment of Copanlisib/Rituximab in patients with MZL in need of treatment, who have failed or are not eligible for local therapy or relapsed after local or systemic therapy. For efficacy the rate of complete remissions (according to the GELA criteria for gastric MALT or to the Cheson 2007 criteria for non-gastric extranodal, nodal and splenic MZL) after induction therapy will be primarily analysed. For toxicity treatment associated adverse events, quality of life and cumulative incidence of secondary malignancies will be documented.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

* Confirmed CD20 positive MALT Lymphoma de novo or relapsed following or being not eligible for local therapy (including surgery, radiotherapy) and antibiotics for H. pylori-positive gastric lymphoma arisen at any extranodal site OR
* Confirmed CD20 positive de novo or relapsed splenic MZL following or not being eligible for local therapy (including surgery and antiviral therapy for Hepatitis C Virus) with symptomatic disease OR
* Confirmed CD20 positive de novo or relapsed nodal MZL Tissue diagnostic procedures must be performed within 12 months prior to study entry and have to include diagnostics by a reference pathology center. Biopsy material from an excisional or core biopsy must be submitted for retrospective central confirmation. Tissue samples dated > 12 months prior to informed consent can be accepted only if tissue material is available for retrospective confirmation, if there is no clinical indication for transformation of disease, and if the request for additional biopsy would be unethical treatment of the patient.

In patients with splenic MZL without splenic tissue available for histologic review, the diagnosis may be confirmed by the presence of splenomegaly and typical morphologic and immunophenotypic findings in the blood and bone marrow. Bone marrow (acceptable up to 12 weeks before start of treatment) must be submitted for retrospective central confirmation.

- Patients in need of treatment: For patients with symptomatic splenic, nodal, or non-gastric extranodal MZL disease that is de novo or has relapsed following local therapy (i.e., surgery or radiotherapy) and requires therapy, as assessed by the investigator.

For nodal MZL and extragastric MALT lymphoma:

- At least one bi-dimensionally measurable lesion (≥ 1.5 cm in its largest dimension by CT scan or MRI). Please refer to Appendix C.

For SMZL:

For splenic MZL, an enlarged spleen on CT scan and lymphoma cell infiltration has to be seen in bone marrow and/or peripheral blood. Please refer also to Appendix E.

At least one of the following criteria must be met:

* Bulky progressive or painful splenomegaly
* one of the following symptomatic/progressive cytopenias: Hb < 10 g/dL, or Plat < 80.000 /µL, or neutropenia < 1000/µL, whatever the reason (autoimmune or hypersplenism or bone marrow infiltration)
* SMZL with concomitant hepatitis C infection which has not responded to or has relapsed after Interferon and/or Ribavirin and/or direct antiviral agents (patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA).
* splenectomised patients with rapidly raising lymphocyte counts, development of lymphadenopathy or involvement of extranodal sites if not being eligible for local therapy.

For gastric MALT lymphoma:

For gastric MALT lymphoma, the clinical evidence of the MZL as seen by gastroendoscopy is sufficient. There is no need to show a measurable lesion by CT scan or MRI. Please refer to Appendix D.

Inclusion is possible for patients with:

* H. pylori-negative disease de novo or following or being not eligible for local therapy (i.e., surgery, radiotherapy or antibiotics) or after systemic therapy.
* H. pylori-positive disease that has remained stable, progressed, or relapsed following antibiotic therapy.

Others:

* Age >= 18 years
* Life expectancy >3 months.
* Baseline platelet Count >= 50 x 109/L (if not due to BM infiltration by the lymphoma), absolute neutrophil Count >= 0.75 x 109/L.
* Meet the following pretreatment laboratory criteria at the Screening visit conducted within 28 days of study enrollment (unless due to underlying lymphoma):

  * ASAT (SGOT): <= 3 times the upper limit of institutional laboratory normal value
  * ALAT (SGPT): <= 3 times the upper limit of institutional laboratory normal value
  * Total Bilirubin: <= 2 mg/dL or 2 times the upper limit of institutional laboratory normal value, unless clearly related to the disease (except if due to Gilbert's syndrome)
* GFR ≥ 40 mL/min/1.73 m²
* Negative HIV antibody
* Positive test results for chronic HBV infection (defined as positive HBsAg serology): patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing. Patients who have protective titers of HBsAb after vaccination or prior but cured hepatitis B are eligible.
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing): patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Pregnancy β-HCG negative. For women of child-bearing potential only (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy); serum or urine β-HCG must be negative during screening and at study enrolment visit
* Premenopausal fertile females must agree to use a highly effective method of birth control for the duration of the therapy up to 12 months after end of therapy. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system ( IUS), bilateral tubal occlusion, vasectomised partner or sexual abstinence. Contraception and pregnancy testing are required according the CTFG recommendations (http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf).
* Men must agree not to father a child for the duration of therapy and 6 months after (use of a condom) and must agree to advice a female partner to use a highly effective method of birth control.
* Willingness and ability to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures, and study restrictions.
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, possible side effects, potential risks and discomforts, and other pertinent aspects of study participation.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrolment:

* ECOG performance status ≥ 2
* History of a non-lymphoid malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥1 year prior to study enrollment visit, other Stage 1 or 2 cancer treated with a curative intent and currently in complete remission, for ≥3 years.
* Central nervous system lymphoma, leptomeningeal lymphoma, or histologic evidence of transformation to a high-grade or diffuse large B-cell lymphoma.
* Ongoing immunosuppressive therapy including corticosteroids (exception < 4 weeks administered at a dose equivalent to ≤ 40 mg/day prednisone is allowed)
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of study enrolment visit
* Ongoing drug-induced liver injury, chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cholangitis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
* Ongoing alcohol or drug addiction
* Treatment with any other investigational agent within 30 days or within 5 x the half-life (t1/2) of the investigational product, whichever is longer, or participating in another trial within 30 days prior to entering this study
* Breastfeeding or pregnancy
* Prior treatment with Copanlisib
* Congestive heart failure > New York Heart Association (NYHA) class 2
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months).
* Myocardial infarction less than 6 months before start of test drug
* Uncontrolled arterial hypertension despite optimal medical management
* HbA1c>8.5%
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram (ECG) finding, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject or impair the assessment of study results.
* History of anaphylaxis in association with previous administration of monoclonal antibodies.
* Vaccination with a live vaccine within 28 days prior to start of therapy
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* Non-healing wound, ulcer, or bone fracture
* History or concurrent interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 12 months
  Primary endpoint is the complete response (CR rate (CRR) determined 12 months after start of induction therapy). Patients who progress before 12 months after start of treatment will be treated as CR='NO' and will be included in the calculation of the primary endpoint. No primary endpoint will be determined for patients who withdraw.

SECONDARY OUTCOMES:
Response rate | 12 months
  The response rates (complete response (CR), partial response (PR)) and overall response rate (CR or PR) are evaluated 4 weeks after the end of induction treatment and 12 months after start of treatment.
Best response | 8.5 years
  Best response is determined in the time interval from the start of induction therapy to end of follow-up.
Time to best response | 8.5 years
  Time to best response is defined as the time from the start of induction to best response the patient achieves (CR, PR).
Time to first response | 12 months
  Time to first response is defined as the time from the start of induction to first response (CR, PR).
Progressioin free survival (PFS) | 12 months
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
Time to Treatment failure (TTF) | 8.5 years
  Time to treatment failure (TTF) is defined as the time of registration to discontinuation of therapy for any reason including death from any cause, progression, toxicity or add-on of new anti-cancer therapy. Patients alive without treatment failure are censored at the latest tumor assessment date.
Duration of Response (DR) | 8.5 years
  Duration of response as defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
Cause specific survival (CSS) | 8.5 years
  Cause specific survival is defined as the period from the induction registration to death from lymphoma or lymphoma related cause; death unrelated to MZL is considered as a competing event.
Overall survival (OS) | 8.5 years
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
Quality of life during induction and maintenance therapy | 8.5 years
  Quality of life will be measured by the FACTLym before start of treatment, during induction and maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Buske, MD, Principal Investigator — University Hospital of Ulm
Locations (18):
- Med. Uni Wien AKH, Klinische Abteilung für Onkologie, Innere Medizin I, Vienna, Austria
- Germany (17):
  - St. Josef-Hospital, Medizinische Klinik I, Bochum
  - Johanniter GmbH, Johanniter-Krankenhaus, Bonn
  - ÜBAG MVZ Dr. Vehling-Kaiser GmbH Dingolfing, Dingolfing
  - Kath. Karl-Leisner-Klinikum gGmbH, Betriebsstätte Wilhelm-Anton-Hospital, Goch
  - MVZ Goslar, MVZ Onkologische Kooperation Harz, Goslar
  - Universitätsklinikum Halle, Klinik und Poliklinik für Innere Medizin, Halle
  - Rotes Kreuz Krankenhaus, Klinik für Interdisziplinäre Onkologie, Kassel
  - ÜBAG MVZ Dr. Vehling-Kaiser GmbH, Landshut
  - Gemeinschaftspraxis, Fachärzte für Innere Medizin, Mannheim
  - Universitätsmedizin Mannheim, III. Medizinische Klinik, Mannheim
  - Kliniken Ostalb Stauferklinikum Schwäbisch Gmünd, Zentrum für Innere Medizin, Mutlangen
  - Klinikum der Universität München, Medizinische Klinik und Poliklinik III, München
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Universitätsklinik PIUS Hospital, Innere Medizin, Oldenburg
  - Elblandkliniken Stiftung & Co. KG, Innere Medizin II, Riesa
  - Universitätsmedizin Rostock, Rostock
  - University Hospital Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grunenberg A, Kaiser LM, Woelfle S, Schmelzle B, Viardot A, Moller P, Barth TFE, Muche R, Dreyhaupt J, Raderer M, Kiesewetter B, Buske C. A phase II study of the PI3K inhibitor copanlisib in combination with the anti-CD20 monoclonal antibody rituximab for patients with marginal zone lymphoma: treatment rationale and protocol design of the COUP-1 trial. BMC Cancer. 2021 Jun 29;21(1):749. doi: 10.1186/s12885-021-08464-6. PMID 34187401